CLINICAL TRIAL: NCT01579955
Title: Non-Interventional Study of NovoSeven® Used in Patients With Haemophilia A and B With Inhibitors Under Normal Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7-1947
Record Dates: First submitted 2012-04-11; First posted 2012-04-18 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- eptacog alpha users
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Prescription of eptacog alpha at the discretion of the physician

SUMMARY:
This study is conducted in Japan. The aim of this non-interventional study is to investigate the safety and effectiveness of treatment with eptacog alpha (NovoSeven®) under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haemophilia A and B with inhibitors who received eptacog alpha (NovoSeven®) as treatment

Exclusion Criteria:

* Patients who was not deemed to be appropriate to the treatment of eptacog alpha (NovoSeven®)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia A and B with inhibitors who received NovoSeven® (eptacog alpha)
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 1999-03-10 (Actual); Primary Completion 2010-03-09 (Actual); Study Completion 2010-03-09 (Actual)

PRIMARY OUTCOMES:
Percentage of bleed treatments resulting in effective bleed resolution: Markedly effective, effective, moderate or ineffective | Year 1
Percentage of bleed treatments resulting in effective bleed resolution: Markedly effective, effective, moderate or ineffective | Year 10

SECONDARY OUTCOMES:
Number of adverse events (AEs), including serious adverse events (SAEs) | Baseline, every 1 year, Year 10

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com